CLINICAL TRIAL: NCT02842034
Title: A Randomized Double-blind Controlled Study of Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Negative Symptoms in Schizophrenia Patients.
Brief Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Negative Symptoms in Schizophrenia Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rTMS-negative symptoms
Record Dates: First submitted 2016-06-20; First posted 2016-07-22 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; rTMS
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Active Comparator): Active treatment will be delivered at an intensity that is 120% of the resting motor threshold (RMT). Stimulation will be delivered at 10 Hz with 60 stimulation trains of 50 stimuli each (i.e., 3000 stimuli) and an intertrain interval of 10 sec. Treatment will be applied in sequential order to the dorsomedial prefrontal cortices (DMPFC).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using the same stimulation parameters and at the same site of active treatment, but the coil will be reversed. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Stimulate the dorsomedial prefrontal cortex for 4 weeks.

SUMMARY:
This study is to determine whether high frequency repetitive transcranial magnetic stimulation (rTMS) is effective in the treatment of negative symptoms in schizophrenia patients

DETAILED DESCRIPTION:
The principal objective of this trial is to investigate the effect of high frequency rTMS on negative symptoms in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of schizophrenia according to DSM-IV；
* 18～55 years old；
* schizophrenic illness duration longer than one year;
* The sum of negative scores in the range Positive and negative symptom score (PANSS) must be 20 points or higher, at least one item from the area of negative symptoms (N1-N7) must be ≥ 4 points (at least moderate, clinically significant symptoms), and improvement in negative symptom-sum (measuring by PANSS) must be 10% or lower during the last two weeks before rTMS stimulation.
* Have a stable and consistent drug treatment at least two weeks prior the rTMS treatment;
* Able to adhere to the treatment schedule;
* IQ≥80;
* Dextromanual, normal vision and hearing;
* Signed an informed consent

Exclusion Criteria:

* rTMS contraindications: intracranial metal substance, with heart pacemakers and cochlear implants, intracranial pressure;
* Acute risk of suicide and impulse；
* patients to be diagnosed according to DSM-IV for substance abused, development delayed;
* suffering from serious physical disease and can not accept the treatment;
* history of epileptic seizures or the presence of epileptic activity documented on the basis of EEG;
* difficult to maintain the current drug treatment for at least 1 month;
* undergoing ECT or MECT in last 3 months;
* current treatment with anticonvulsant acting drugs such as anticonvulsants, benzodiazepines.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in clinical improvement of negative symptoms (Scale for Assessment of Negative Symptoms [SANS], and Positive and Negative Syndrome Scale [PANSS] negative symptoms subscale) | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale [PANSS] positive symptoms subscale | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in Calgary Depression Scale for Schizophrenia [CDSS] | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in clinical global impression [CGI] | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in WHO Disability Assessment Schedule 2.0 [WHODAS 2.0] | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in Simpson-Angus Scale [SAS] | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in Clinician Rated Dimensions of Psychosis Symptom [CRDPS] | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)

OTHER OUTCOMES:
Change from baseline in Letter-Number Span | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in Wechsler Working Memory | 3 times (Before treatment,immediately after treatment,4 weeks after treatment)
Change from baseline in Resting-state functional MRI:TR=2000 ms，TE=35 ms，FA=90，Matrix =64×64，Nex=1，FOV=256 mm，thickness=4 mm，Gap=0,scanning 33 slices。 | 2 times (Before treatment,immediately after treatment)
Change from baseline in diffusion tensor imaging (DTI):TR=8500,TE=87, matrix size=64×64, FOV=230, slices thickness = 3 mm, diff directions=30,scanning 46 slices | 2 times (Before treatment,immediately after treatment)
Change from baseline in Magnetic Resonance Spectroscopy (MRS) of DMPFC | 2 times (Before treatment,immediately after treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China